CLINICAL TRIAL: NCT01755156
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, and Efficacy of the Addition of MK-3102 to Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Therapy
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of the Addition of Omarigliptin (MK-3102) to Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Therapy (MK-3102-024)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3102-024; 2012-003670-11 (EudraCT Number)
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; glimepiride; Insulin Glargine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omarigliptin (Phase A) → Omarigliptin (Phase B) (Experimental): Phase A: Omarigliptin 25 mg capsule administered orally once weekly for 24 weeks. Phase B: Omarigliptin 25 mg capsule administered orally once weekly and matching placebo to glimepiride tablet/capsule administered orally once daily for 80 weeks. Participants will continue pre-study metformin throughout the duration of the study. If necessary, rescue therapy may be initiated (open-label glimepiride during Phase A and insulin glargine during Phase B).
  Interventions: Drug: Omarigliptin; Drug: Matching placebo to glimepiride; Drug: Insulin glargine; Drug: Metformin
- Placebo to omarigliptin (Phase A) → Glimepiride (Phase B) (Placebo Comparator): Phase A: matching placebo to omarigliptin orally once a week for 24 weeks. Phase B: Matching placebo to omarigliptin capsule administered orally once weekly and glimepiride 1 or 2 mg tablet/capsule administered orally once daily (titrated up to 6 mg daily) for 80 weeks. Participants will continue pre-study metformin throughout the duration of the study. If necessary, rescue therapy may be initiated (open-label glimepiride during Phase A and insulin glargine during Phase B).
  Interventions: Drug: Matching placebo to omarigliptin; Drug: Glimepiride; Drug: Insulin glargine; Drug: Metformin

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin 25 mg capsule administered orally once weekly (preferably on the same day of each week)
  Other Names: MK-3102
  Arms: Omarigliptin (Phase A) → Omarigliptin (Phase B)
Drug: Matching placebo to omarigliptin — Matching placebo to omarigliptin capsule administered orally once weekly (preferably on the same day of each week)
  Arms: Placebo to omarigliptin (Phase A) → Glimepiride (Phase B)
Drug: Glimepiride — Glimepiride 1 or 2 mg tablet/capsule administered orally once daily and up-titrated to a maximum dose of 6 mg daily. Participants rescued with open-label glimepiride during Phase A will not receive glimepiride or matching placebo to glimepiride during Phase B.
  Other Names: Amaryl®
  Arms: Placebo to omarigliptin (Phase A) → Glimepiride (Phase B)
Drug: Matching placebo to glimepiride — Matching placebo to glimepiride tablet/capsule administered orally once daily and up-titrated to a mock maximum dose of 6 mg daily. Participants rescued with open-label glimepiride during Phase A will not receive glimepiride or matching placebo to glimepiride during Phase B.
  Arms: Omarigliptin (Phase A) → Omarigliptin (Phase B)
Drug: Insulin glargine — During Phase B of the study, participants who received a maximum up-titration of open-label glimepiride or blinded glimepiride/matching placebo to glimepiride, may be rescued with open-label insulin glargine.
  Other Names: Lantus
Drug: Metformin — Participants continue stable pre-study dose of metformin tablet(s) administered orally (>= 1500 mg daily) throughout the study.
  Other Names: Fortamet®; Glucophage®; Glucophage® XR; Glumetza®; Riomet®; Metgluco®; Glycoran®

SUMMARY:
The purpose of this study is to assess the safety and efficacy of omarigliptin compared to placebo in participants with inadequate glycemic control on metformin monotherapy. The primary hypothesis is that after 24 weeks, the addition of treatment with omarigliptin provides greater reduction in hemoglobin A1c (A1C) than placebo.

DETAILED DESCRIPTION:
Participants received blinded omarigliptin or matching placebo to omarigliptin for 104 weeks. During the first 24 weeks (Phase A) they did not receive any other blinded study medication. In Phase B (subsequent 80 weeks), participants who did not initiate glycemic rescue in Phase A received additional blinded study medication: participants in the omarigliptin group received placebo to glimepiride and participants in the placebo group received glimepiride.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus
* Currently on a stable dose of metformin monotherapy (>=1500 mg per day) for at least 12 weeks prior to study participation
* Male, or female who is not of reproductive potential or if of reproductive potential agrees to abstain from heterosexual activity or use (or have their partner use) acceptable contraception to prevent pregnancy during the study and for 21 days after the last dose of study drug

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* Has been treated with any antihyperglycemic agent (AHA) other than the protocol-required metformin within 12 weeks prior to study participation or with omarigliptin at any time prior to signing informed consent
* History of hypersensitivity to a dipeptidyl peptidase IV (DPP-4) inhibitor
* History of intolerance, hypersensitivity, or any other contraindication to metformin, glimepiride, or insulin glargine
* Is on a weight loss program and is not in the maintenance phase or has been on a weight loss medication in the past 6 months or has undergone bariatric surgery within 12 months prior to study participation
* Has undergone a surgical procedure within 4 weeks of study participation or has planned major surgery during the study
* Is on or likely to require treatment for >=2 consecutive weeks or repeated courses of corticosteroids (inhaled, nasal and topical corticosteroids are permitted)
* Currently being treated for hyperthyroidism or is on thyroid hormone replacement therapy and has not been on a stable dose for at least 6 weeks
* Is expecting to undergo hormonal therapy in preparation to donate eggs during the period of the trial, including 21 days after the last dose of blinded study medication
* History of active liver disease (other than non-alcoholic steatosis) including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Human immunodeficiency virus (HIV)
* New or worsening signs or symptoms of coronary heart disease or congestive heart failure within the past 3 months, or myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous transluminal coronary angioplasty, stroke, or transient ischemic attacks in the past 3 months
* Poorly controlled hypertension
* History of malignancy <=5 years prior to study participation, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Positive urine pregnancy test
* Pregnant or breastfeeding, or is expecting to conceive during the study including 21 days following the last dose of blinded study drug
* User of recreational or illicit drugs or has had a recent history of drug abuse
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking
* Has donated blood products or has had phlebotomy of >300 mL within 8 weeks of study participation, or intends to donate blood products within the projected duration of the trial or has received, or is anticipated to receive, blood products within 12 weeks of study participation or within the projected duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2013-01-11 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Shankar RR, Inzucchi SE, Scarabello V, Gantz I, Kaufman KD, Lai E, Ceesay P, Suryawanshi S, Engel SS. A randomized clinical trial evaluating the efficacy and safety of the once-weekly dipeptidyl peptidase-4 inhibitor omarigliptin in patients with type 2 diabetes inadequately controlled on metformin monotherapy. Curr Med Res Opin. 2017 Oct;33(10):1853-1860. doi: 10.1080/03007995.2017.1335637. Epub 2017 Jun 23. PMID 28547998

RESULTS

PARTICIPANT FLOW:
Groups:
- Omarigliptin (Phase A) → Omarigliptin (Phase B): Phase A: Omarigliptin 25 mg capsule administered orally once weekly for 24 weeks. Phase B: Omarigliptin 25 mg capsule administered orally once weekly and matching placebo to glimepiride tablet/capsule administered orally once daily for 80 weeks.
- Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B): Phase A: matching placebo to omarigliptin orally once a week for 24 weeks. Phase B: Matching placebo to omarigliptin capsule administered orally once weekly and glimepiride 1 or 2 mg tablet/capsule administered orally once daily (titrated up to 6 mg daily) for 80 weeks.
Period: Phase A (Weeks 0-24)
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Started | 201 | 201
Completed | 184 | 177
Not Completed | 17 | 24
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 5 | 3
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Creatinine or eGFR Discon. Criteria | 0 | 2
Not completed — Need for Excluded Med. Discon. Criteria | 1 | 1
Period: Phase B (Weeks 24-104)
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Started | 183 (1 participant who completed Phase A did not continue to Phase B.) | 177
Completed | 144 | 141
Not Completed | 39 | 36
Not completed — Lost to Follow-up | 12 | 5
Not completed — Withdrawal by Subject | 27 | 31

BASELINE CHARACTERISTICS:
Groups:
- Omarigliptin (Phase A): Phase A: Omarigliptin 25 mg capsule orally once a week for 24 weeks.
- Placebo to Omarigliptin (Phase A): Phase A: Matching placebo to omarigliptin capsule administered orally once weekly for 24 weeks
- Total: Total of all reporting groups
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A) | Total
Number analyzed (Participants) | 201 | 201 | 402
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (8.1) | 56.8 (9.1) | 57.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 99 | 199
  Male | 101 | 102 | 203
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent] | 8.06 (0.87) | 8.02 (0.89) | 8.04 (0.88)
2-hour post-meal glucose (2-hr PMG) [Mean (Standard Deviation); unit: mg/dL] — Omarigliptin (Phase A), n=192; Placebo to omarigliptin (Phase A), n=193; Total, n=385
  mg/dL | 240.2 (60.5) | 236.0 (59.9) | 238.1 (60.2)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 168.8 (37.6) | 168.6 (37.2) | 168.7 (37.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (A1C) at Week 24 (Phase A)
Description: A1C is measured as a percent. Change from baseline in A1C at Week 24 was analyzed using a constrained longitudinal data analysis (cLDA) method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, time, and the interaction of time by treatment.
Time Frame: Baseline and Week 24
Population: Full analysis set population included all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 201 | 201
Percent | -0.54 [-0.69 to -0.40] | 0.00 [-0.14 to 0.15]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p < 0.001, cLDA; Based on a cLDA method with a restriction of the same baseline mean; Difference in least squares means = -0.55, 95% CI 2-sided [-0.75 to -0.34]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (Phase A+B)
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. Presented data exclude data after glycemic rescue.
Time Frame: Up to 107 weeks
Population: All participants as treated population included all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 65.7 | 65.2
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) → Omarigliptin (Phase B) vs Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B); Test type: Superiority or Other; Difference in % = 0.5, 95% CI 2-sided [-8.8 to 9.8] — Based on Miettinen & Nurminen method. The 95% CI was computed only for those endpoints with at least 4 participants having events in 1 or more treatment groups

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event (Phase A+B)
Description: as for outcome 2
Time Frame: Up to 104 weeks
Population: All participants as treated population included all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 2.0 | 4.5
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) → Omarigliptin (Phase B) vs Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B); Test type: Superiority or Other; Difference in % = -2.5, 95% CI 2-sided [-6.6 to 1.1] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event Which Were Included Under the System Order Class of Investigations (Phase A+B)
Description: The following laboratory parameters were included: blood chemistry, hematology, electrocardiograms, lipids, body weight, and vital signs.
Time Frame: Up to 104 weeks
Population: All participants as treated population included all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 21.9 | 17.4
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) → Omarigliptin (Phase B) vs Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B); Test type: Superiority or Other; Difference in % = 4.5, 95% CI 2-sided [-3.3 to 12.3]

5. Secondary Outcome: Change From Baseline in 2-hour Post-meal Glucose (PMG) at Week 24 (Phase A)
Description: Change from baseline in 2-hour PMG at Week 24 was analyzed using cLDA method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, time, and the interaction of time by treatment.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 195 | 199
mg/dL | -26.8 [-34.8 to -18.7] | -12.2 [-20.7 to -3.8]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.011, cLDA; Based on a cLDA method with a restriction of the same baseline mean; Difference in % = -14.5, 95% CI 2-sided [-25.6 to -3.4]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 (Phase A)
Description: Change from baseline in FPG at Week 24 was analyzed using cLDA method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, time, and the interaction of time by treatment.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 201 | 201
mg/dL | -10.7 [-16.0 to -5.5] | -1.2 [-6.6 to 4.1]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.010, cLDA; Based on a cLDA method with a restriction of the same baseline mean; Difference in least squares means = -9.5, 95% CI 2-sided [-16.7 to -2.3]

7. Secondary Outcome: Change From Baseline in A1C at Week 104 (Phase A+B)
Description: A1C is measured as a percent. Change from baseline in A1C at Week 104 was analyzed using cLDA method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, time, and the interaction of time by treatment.
Time Frame: Baseline and Week 104
Population: Full analysis set population included all randomized participants who received at least one dose of study medication and had a baseline measurement or a post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
Percent | -0.42 [-0.59 to -0.25] | -0.51 [-0.68 to -0.34]

8. Secondary Outcome: Change From Baseline in FPG at Week 104 (Phase A+B)
Description: Change from baseline in FPG at Week 104 was analyzed using cLDA method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, time, and the interaction of time by treatment.
Time Frame: Baseline and Week 104
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
mg/dL | -7.8 [-14.4 to -1.3] | -18.2 [-24.7 to -11.7]

9. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <7.0% After 24 Weeks of Treatment (Phase A)
Description: Percentage of participants attaining A1C glycemic goals of <7.0% (53 mmol/mol) after 24 weeks of treatment estimated using standard multiple imputation techniques.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 38.0 [31.3 to 45.1] | 18.8 [13.9 to 25.0]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen method; Between-group rate difference (%) = 19.2, 95% CI 2-sided [10.1 to 28.0]

10. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <6.5% After 24 Weeks of Treatment (Phase A)
Description: Percentage of participants attaining A1C glycemic goals of <6.5% (48 mmol/mol) after 24 weeks of treatment estimated using standard multiple imputation techniques.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 10.6 [6.8 to 16.2] | 6.4 [3.6 to 11.2]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.164, Miettinen & Nurminen method; Between-group rate difference (%) = 4.2, 95% CI 2-sided [-1.8 to 10.5]

11. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <7% After 104 Weeks of Treatment (Phase A+B)
Description: Percentage of participants attaining A1C glycemic goals of <7.0% (53 mmol/mol) after 104 weeks of treatment estimated using standard multiple imputation techniques.
Time Frame: 104 weeks
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 32.2 [25.7 to 39.5] | 39.0 [31.7 to 46.8]

12. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <6.5% After 104 Weeks of Treatment (Phase A+B)
Description: Percentage of participants attaining A1C glycemic goals of <6.5% (48 mmol/mol) after 104 weeks of treatment estimated using standard multiple imputation techniques.
Time Frame: 104 weeks
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 13.7 [9.4 to 19.6] | 17.9 [12.5 to 24.8]

13. Secondary Outcome: Change From Baseline in PMG Total Area Under the Plasma Concentration Time Curve (AUC) at Week 24 (Phase A)
Description: Change from baseline in PMG total AUC at Week 24 based on a cLDA model including terms for treatment, time, and the interaction of time by treatment. Plasma glucose levels were measured before the meal (0 minutes), and at 60 and 120 minutes after the meal.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg*h/dL
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 195 | 198
mg*h/dL | -46.4 [-58.7 to -34.1] | -18.6 [-31.5 to -5.7]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.001, cLDA; Based on a cLDA method with a restriction of the same baseline mean; Difference in least squares means = -27.8, 95% CI 2-sided [-44.8 to -10.8]

14. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 24 (Phase A)
Description: Change from baseline in fasting insulin at Week 24 based on a cLDA model including terms for treatment, time, and the interaction of time by treatment.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: micro International Unit (μIU)/mL
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 200 | 200
micro International Unit (μIU)/mL | 1.8 [-0.6 to 4.2] | -1.9 [-4.3 to 0.5]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.025, cLDA; Based on a cLDA method with a restriction of the same baseline mean; Difference in least squares means = 3.7, 95% CI 2-sided [0.5 to 6.9]

15. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 104 (Phase A+B)
Description: Change from baseline in fasting insulin at Week 104 based on a cLDA model including terms for treatment, time, and the interaction of time by treatment.
Time Frame: Baseline and Week 104
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: μIU/mL
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 200
μIU/mL | 1.2 [-1.9 to 4.2] | 1.8 [-1.2 to 4.8]

16. Secondary Outcome: Kaplan-Meier Estimate of Cumulative Incidence of Participants Requiring Glycemic Rescue Therapy by 24 Weeks (Phase A)
Description: Participants who did not meet progressively stricter glycemic criteria in Phase A had rescue initiated with open-label glimepiride.
Time Frame: Up to 24 weeks
Population: All participants randomized population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 8.5 [5.3 to 13.6] | 9.7 [6.2 to 15.0]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.654, Log Rank; Kaplan-Meier difference % = -1.2, 95% CI 2-sided [-7.0 to 4.7]

17. Secondary Outcome: Kaplan-Meier Estimate of Cumulative Incidence of Participants Requiring Glycemic Rescue Therapy by 104 Weeks (Phase A+B)
Description: Participants who did not meet progressively stricter glycemic criteria in Phase A had rescue initiated with open-label glimepiride. If during Phase B participants on open-label glimepiride or blinded glimepiride/glimepiride matching placebo needed rescue after maximum up-titration, then insulin glargine was initiated and the dose of open-label glimepiride or blinded glimepiride/glimepiride-matching placebo was discontinued.
Time Frame: Up to 104 weeks
Population: All participants randomized population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 20.2 [14.9 to 27.1] | 16.2 [11.5 to 22.7]

18. Secondary Outcome: Percentage of Participants Requiring Glycemic Rescue Therapy at or Before Week 24 (Phase A)
Description: Data presented are a cumulative incidence of participants with glycemic rescue by Week 24.
Time Frame: Up to 24 weeks
Population: All participants randomized population.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 8.0 [5.3 to 13.6] | 9.0 [6.2 to 15.0]

19. Secondary Outcome: Percentage of Participants Requiring Glycemic Rescue Therapy at or Before Week 104 (Phase A+B)
Description: Data presented are a cumulative incidence of participants with glycemic rescue by Week 104.
Time Frame: Up to 104 weeks
Population: All participants randomized population.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Number analyzed (Participants) | 201 | 201
Percentage of participants | 17.4 | 13.9

ADVERSE EVENTS:
Time Frame: Up to 107 weeks (treatment period + 21-day follow-up)
Description: APaT population consists of all randomized participants who took at least 1 dose of study drug. Serious adverse events (SAEs) include data after glycemic rescue; non-serious adverse events exclude data after glycemic rescue. The AEs reported in the (Phase A) → (Phase B) columns are a total of the AEs (SAEs) that occurred in Phases A and B.
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A) | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B)
Serious Adverse Events (participants affected / at risk) | 5/201 | 10/201 | 12/201 | 18/201
Other Adverse Events (participants affected / at risk) | 27/201 | 17/201 | 53/201 | 58/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (Phase A) (N=201) | Placebo to Omarigliptin (Phase A) (N=201) | Omarigliptin (Phase A) → Omarigliptin (Phase B) (N=201) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B) (N=201)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (Phase A) (N=201) | Placebo to Omarigliptin (Phase A) (N=201) | Omarigliptin (Phase A) → Omarigliptin (Phase B) (N=201) | Placebo to Omarigliptin (Phase A) → Glimepiride (Phase B) (N=201)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1) | 11 (12) | 7 (7)
Blood glucose increased (Investigations) | 9 (9) | 7 (10) | 14 (16) | 10 (14)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (13) | 5 (8) | 17 (43) | 32 (112)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 11 (12) | 8 (9)
Headache (Nervous system disorders) | 5 (5) | 5 (5) | 8 (8) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.